CLINICAL TRIAL: NCT04089384
Title: Effectiveness of Integrative and Complementary Practice in Health as a Strategy in Obesity Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Pernambuco (Other)
Responsible Party: Principal Investigator, Cicero Jonas Rodrigues Benjamim, Principal Investigator, University of Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPernambuco11-09
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Obesity; Weight Loss
Keywords: Obesity; Auriculotherapy; Weight Loss; Nutrition Therapy
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: All patients selected for the research will be interviewed by the same Nutritionist, responsible for the anthropometric assessment, who will use a specific questionnaire to record the personal, socioeconomic and lifestyle information of the patients. A. Control Group: Patients in this group will receive an individualized eating plan every 15 days and a marked micropore. B. Auriculotherapy group: will receive individualized eating plan every 15 days and will undergo 12 auriculotherapy sessions, 1 per week, lasting 5 to 10 minutes for each session, will be compressed by mustard seed in the following points; mouth, stomach, anxiety, hunger and Shen Men. C. Placebo group: will receive individualized eating plan every 15 days and will undergo 12 auriculotherapy sessions, similar to the auriculotherapy group, but the applications will be in sham points, points not indicative for the proposed treatment, wrist and outer ear points.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Other): Will receive individualized dietary plan - alimentary reeducation and micropore containing a point made with a black gel pen that will be placed in the ear
  Interventions: Other: Control Group
- Auriculotherapy Group (Active Comparator): Will receive individualized diet plan - diet reeducation and auricular therapy method with strategic points for obesity
  Interventions: Other: Auriculotherapy Group
- Placebo group (Placebo Comparator): Will receive individualized diet plan - diet reeducation and sham points, points not indicative for the proposed treatment
  Interventions: Other: Placebo group

INTERVENTIONS:
Other: Control Group — Will receive individualized dietary plan - alimentary reeducation and micropore containing a point made with a black gel pen that will be placed in the ear
  Arms: Control Group
Other: Auriculotherapy Group — Will receive individualized diet plan - diet reeducation and auricular therapy method with strategic points for obesity
  Arms: Auriculotherapy Group
Other: Placebo group — Will receive individualized diet plan - diet reeducation and sham points, points not indicative for the proposed treatment).
  Arms: Placebo group

SUMMARY:
Obesity is highlighted, pointed as a disease that has been increasingly affecting individuals and becoming an epidemic in recent decades, but auriculotherapy has been shown to contribute to the treatment of this disease.The objective of this study was to evaluate the therapeutic efficacy of auriculotherapy associated with dietary education in reducing weight in obese patients. This is a simple-blind Randomized Clinical Trial.

DETAILED DESCRIPTION:
Considering the low cost, benefits and applicability of auriculotherapy in the integral care of the individual, as well as the remaining gap regarding studies involving the practice of auriculotherapy in obese patients with a representative sample, this study will be conducted with The objective of this study was to evaluate the therapeutic efficacy of auriculotherapy associated with dietary education in reducing weight in obese patients.

The study will be performed at the nutrition laboratory III of the University of Pernambuco (UPE) Petrolina campus, with users previously diagnosed with obesity. This is a simple-blind Randomized Clinical Trial, with 3 groups: control group (will receive individualized dietary plan - alimentary reeducation and micropore containing a point made with a black gel pen that will be placed in the ear); auriculotherapy group (will receive individualized diet plan - diet reeducation and auricular therapy method with strategic points for obesity) and placebo group (will receive individualized diet plan - diet reeducation and sham points, points not indicative for the proposed treatment).

Will be included in the study all adult patients of both sexes in the age of 20 years complete for 44 incomplete years, who meet the eligibility criteria.

- Inclusion criteria: All adult patients seeking treatment for weight loss in August 2019 at the UPE and who agree to participate in the study by signing the Informed Consent Form (ICF). - Exclusion criteria: Pregnant women, patients who are treated with obesity secondary to some pathology and need previous treatment for hormonal control, or have not properly completed or signed the informed consent form.

The sample size was estimated by the EPI INFO software, version 3.5.1. For the calculation it was considered that 20% of adults are obese and 30% have adequate nutritional status, assuming a relative risk of 1.5 to be obese, for a significance level of 95% (1-alpha) and a power value. 80% (1-alpha) with the ratio of unexposed / exposed being 1: 1. . The estimated value of the sample was 36 adults in each group, and the total sample 108, adding 10% in each group to compensate for any losses, resulted in a final sample of 120 individuals, with no 40 participants per group.

Randomization will be performed near the beginning of the intervention by a researcher not involved in the study using the Epitable application's random number table from the EPI-INFO software. The codes that will define which group the recruited obese patients (Control group, auriculotherapy or placebo) will belong to will be placed in opaque envelopes and sealed by one of the researchers who will not be involved in opening them, and upon recruitment, will be opened by the research assistant, who will register the patients, following the sequence of the drawn envelopes.

:

ELIGIBILITY:
Inclusion Criteria:

* Obesity
* Body Mass Index: > 29,9kg/m²

Exclusion Criteria:

* Pregnant women
* Patients with treatment secondary
* Need previous treatment for hormonal control
* Have not properly completed or signed the informed consent form

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 12 weeks
  Weight loss will be verified by means of kilogram (kg)
Abdominal circumferece | 12 weeks
  Will be measured by the abdominal circumference measured in centimeters (cm)
Cardiovascular risk | 12 weeks
  The waist circumference in centimeters (cm) will be used to assess the decrease in cardiovascular risk, considering the cutoff points of the world health organization.
  Men -Increased ≥ 94 cm; Substantially increased ≥ 102cm.
  Woman - Increased ≥ 80 cm; Substantially increased ≥ 88cm.
Height | 12 weeks
  The height measured shall be taken to the extent of centimeters (cm)
Body Max Index | 12 weeks
  Body Mass Index (BMI) will be evaluated from weight (kg) and height (m) using the formula (kg/ m²).

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Galdino, Study Chair — University of Pernambuco; Andrea Sotero, phD, Study Director — University of Pernambuco

IPD SHARING:
Plan to Share IPD: Undecided